CLINICAL TRIAL: NCT00182871
Title: Testosterone Effects on Bone and Frailty in Men With Osteoporosis
Brief Title: Testosterone Effects on Bone and Frailty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AG0043; R01AG018887 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: Aging; Frailty; Osteoporosis
Keywords: geriatric medicine; hormone therapy; HT; andropause
MeSH Terms: conditions — Frailty; Osteoporosis | interventions — Testosterone

INTERVENTIONS:
Drug: testosterone

SUMMARY:
The purpose of this study is to assess the effects of testosterone replacement on bone density, muscle strength, physical performance, quality of life and prostate symptoms in men selected for low bone mineral density or fracture and some aspect of frailty.

DETAILED DESCRIPTION:
The hypothesis being tested is that testosterone supplementation can increase bone mineral density and specific parameters of frailty in older men with osteoporosis and characteristics of frailty. One hundred and eighty men, age 60 years and older, who have sustained a hip fracture or other fragility fracture following mild to moderate trauma (such as a fall from standing height) in the previous 5 years or who have low femoral neck bone mineral density plus a component of frailty (weight loss, perception of exhaustion, physical strength, physical activity level and walking time) will be randomly assigned to receive either testosterone or placebo, delivered by topical gel applied daily, in a two year double-blind study.

Bone mineral density (BMD) by dual x-ray absorptiometry (DXA), will be performed at baseline and yearly to assess changes in BMD. Blood and urine samples will be collected at baseline and yearly; these tests will be correlated to changes in BMD.

To determine the effects of testosterone on frailty, strength of the upper and lower extremities will be measured every 6 months using the hand-held dynamometer and sitting leg press, respectively. Changes in lean body mass and percent body fat will be measured by total body DXA at baseline, 6 months and then annually. In addition, physical performance, emotional and sexual function, and disability will be assessed also.

The safety of testosterone supplementation on prostate and cardiovascular parameters will also be monitored; participants will be screened for prostate cancer at baseline, 6 months then yearly for 2 years. Fasting lipoprotein levels will be measured yearly while on testosterone replacement, and cardiovascular specific adverse effects such as angina, myocardial infarction, stroke and sudden death will be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Men over age 60 years who have sustained a femoral fracture in the preceding 3 years
* Total testosterone levels below 375 ng/dl or bioavailable testosterone levels at least 1.5 SD lower than the young adult mean
* Able to come or be brought to the University of Connecticut Health Center (UCHC) for outpatient visits

Exclusion Criteria:

* Prostate specific antigen level over 4.0 ng/dl or the history of prostate cancer
* Disease of bone metabolism (i.e., Paget's disease, osteomalacia, hyperparathyroidism)
* History of pituitary disease
* History of sleep apnea
* Consumption of more than 3 alcoholic drinks/day
* Use of androgen, estrogen, or DHEA in the preceding year
* Use of antiresorptive agents such as calcitonin or bisphosphonates
* Metastatic or advanced cancer
* Current chemotherapy or radiation treatment
* Plans to move in the next three years
* Advanced liver or renal disease such that the subjects is unlikely to complete the three year intervention
* Hemaglobin >16.5 g/dl
* Bilateral hip replacement or repair

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2001-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Bone density and strength

SECONDARY OUTCOMES:
Physical performance
quality of life
cognition
lipids
prostate specific antigen
prostate symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kenny, MD, Principal Investigator — Center on Aging, University of Connecticut Health Center
Locations (1):
- Center on Aging, University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] Tenover JL. Testosterone and the aging male. J Androl. 1997 Mar-Apr;18(2):103-6. PMID 9154502
- [Background] Morley JE, Perry HM 3rd, Kaiser FE, Kraenzle D, Jensen J, Houston K, Mattammal M, Perry HM Jr. Effects of testosterone replacement therapy in old hypogonadal males: a preliminary study. J Am Geriatr Soc. 1993 Feb;41(2):149-52. doi: 10.1111/j.1532-5415.1993.tb02049.x. PMID 8426037
- [Background] Snyder PJ, Peachey H, Hannoush P, Berlin JA, Loh L, Holmes JH, Dlewati A, Staley J, Santanna J, Kapoor SC, Attie MF, Haddad JG Jr, Strom BL. Effect of testosterone treatment on bone mineral density in men over 65 years of age. J Clin Endocrinol Metab. 1999 Jun;84(6):1966-72. doi: 10.1210/jcem.84.6.5741. PMID 10372695
- [Background] Kenny AM, Prestwood KM, Gruman CA, Marcello KM, Raisz LG. Effects of transdermal testosterone on bone and muscle in older men with low bioavailable testosterone levels. J Gerontol A Biol Sci Med Sci. 2001 May;56(5):M266-72. doi: 10.1093/gerona/56.5.m266. PMID 11320105
- [Background] Kenny AM, Bellantonio S, Gruman CA, Acosta RD, Prestwood KM. Effects of transdermal testosterone on cognitive function and health perception in older men with low bioavailable testosterone levels. J Gerontol A Biol Sci Med Sci. 2002 May;57(5):M321-5. doi: 10.1093/gerona/57.5.m321. PMID 11983727
- [Background] Kenny AM, Prestwood KM, Gruman CA, Fabregas G, Biskup B, Mansoor G. Effects of transdermal testosterone on lipids and vascular reactivity in older men with low bioavailable testosterone levels. J Gerontol A Biol Sci Med Sci. 2002 Jul;57(7):M460-5. doi: 10.1093/gerona/57.7.m460. PMID 12084809
- [Derived] Kenny AM, Kleppinger A, Annis K, Rathier M, Browner B, Judge JO, McGee D. Effects of transdermal testosterone on bone and muscle in older men with low bioavailable testosterone levels, low bone mass, and physical frailty. J Am Geriatr Soc. 2010 Jun;58(6):1134-43. doi: 10.1111/j.1532-5415.2010.02865.x. PMID 20722847